CLINICAL TRIAL: NCT07287202
Title: An Open-Label Phase 1b/2a Study to Evaluate the Safety and Tolerability of Oral SVG103 (Paxalisib) in Adults With Focal Cortical Dysplasia Type II (FCD-II), Tuberous Sclerosis Complex (TSC) or Hemimegalencephaly (HME), Followed by Long-Term Treatment
Brief Title: Safety, Tolerability, and Pharmacokinetics of SVG103 (Paxalisib) in Focal Cortical Dysplasia Type II (FCD-II), Tuberous Sclerosis Complex (TSC) or Hemimegalencephaly (HME)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sovargen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVG103-001
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Focal Cortical Dysplasia; Tuberous Sclerosis Complex (TSC); Hemimegalencephaly
Keywords: FCD-II; TSC; HME
MeSH Terms: conditions — Focal Cortical Dysplasia; Tuberous Sclerosis; Hemimegalencephaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm1 (Experimental): Drug: SVG103 capsule It will be administered once a day (q.d.) orally.
  Interventions: Drug: SVG103

INTERVENTIONS:
Drug: SVG103 — The study treatment is administered for 3 months during the core phase and for an additional 6 months during the extension phase. Oral, daily, dosage per protocol.
  Other Names: paxalisib

SUMMARY:
This is a multinational, open-label, single-arm trial of adjunctive SVG103 (paxalisib) treatment in adults with FCD-II, TSC, and HME.

DETAILED DESCRIPTION:
This is an open-label, phase 1b/2a study to evaluate safety, tolerability, and pharmacokinetics SVG103 (paxalisib) in 15 patients with Focal Cortical Dysplasia Type II (FCD-II), Tuberous Sclerosis Complex (TSC) or Hemimegalencephaly (HME).

The name of the study drug involved in this study is SVG103 (paxalisib).

The trial consists of two parts: the core phase consists of a 4 week prospective baseline period (D-28~D1) to collect seizure data, followed by a 12-week treatment phase. The extension phase consists of a 24-week treatment period. For participants not continuing in the extension phase, there is a 4-week washout (follow-up) phase.

It is expected that about 15 participants will take part in this research study for up to 9 months as long as there is no serious side effects and disease progression.

"Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved SVG103 (paxalisib) for this specific disease.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants diagnosed with:

   * FCD-II: diagnosis of FCD Type II based on clinical symptoms and confirmed by a positive magnetic resonance imaging (MRI) or histological/pathological analysis of brain tissue, or
   * TSC: diagnosis of TSC by either clinical or genetic diagnostic criteria as documented in the participant's medical record, or
   * HME: Definitive HME confirmed with MRI.
2. Male or female between the ages of 18 and 65 years of age (inclusive).
3. History of failure to control seizures despite at least 2 ASMs at appropriate dosages and duration of treatment.
4. Participants must have experienced at least 8 countable seizures per month for 2 of the 3 months as documented in historical seizure diaries before the baseline period.

6. If participants are on a ketogenic or modified atkins diet, that the regimen can remain unchanged throughout the study, in the opinion of the investigator.

7. Participants with Neurostimulation devices (i.e. Vagus Nerve Stimulation (VNS), Responsive Neuro Stimulation (RNS), Deep Brain Stimulation (DBS) who meet all of the following conditions:

* The device has been implanted for ≥1 year prior to the screening visit.
* The settings must have remained constant for 3 months prior to the screening visit and can remain constant throughout the study, in the opinion of the investigator.
* The battery is expected to last throughout the study. 8. A participant/caregiver or LAR willing to give written informed consent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures.

Key Exclusion Criteria:

1. Clinically significant hepatic, renal, pulmonary, gastrointestinal, neurological (other than epilepsy; HME; TSC; FCD-II), autoimmune, immunological, infections, hematological, malignant conditions that may interfere with or impact the participation in the study or study conduct, as determined but the investigator or sponsor.
2. Immunocompromised participants, defined as acquired immune deficiency syndrome (AIDS), cancer, malnutrition, and certain genetic disorders or undergoing treatment with anticancer drugs, radiation therapy, and stem cell or organ transplant.
3. Participants who have an active central nervous system (CNS) infection, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive as evaluated by brain imaging (magnetic resonance imaging [MRI]).
4. Participants being considered for brain surgery during the study or has undergone brain surgery within 6 months prior to screening visit for epilepsy or any other reason.
5. Participants with HbA1c levels ≥9.0%, or with hyperglycemia or diabetes requiring insulin therapy, or significant uncontrolled hyperglycaemia or diabetes mellitus that would compromise patient safety, as determined by the investigator.
6. Participants with active pneumonitis that are clinically symptomatic.
7. Participants with a history of myocardial infarction or coronary artery disease or clinically significant ECG abnormality.
8. Participants who have clinically significant hepatic, renal and blood laboratory values at baseline period.
9. Participants with known sensitivity or allergy to any component in the investigational product(s) (microcrystalline cellulose, lactose monohydrate, croscarmellose sodium, and colloidal silicon dioxide).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (SAEs), Adverse Drug Reactions (ADRs), TEAEs Leading to Discontinuation and Severity of TEAEs | Up to 36 Weeks
  An adverse event (AE) was any untoward medical occurrence in a clinical study patient, temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event was any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or any other event that requires scientific judgment.

SECONDARY OUTCOMES:
Change from baseline in seizure frequency | Baseline to Core Phase: week 1 to 12 and Baseline to Extension Phase: week 13 to 36
  Assessed by seizure diaries

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred, Melbourne, Victoria